CLINICAL TRIAL: NCT06003647
Title: Educational Intervention Among Informal Caregivers of Person With Dementia in Klang Valley, Malaysia
Brief Title: Educational Intervention Among Informal Caregivers of Person With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Nuraisyah Hani Binti Zulkifley, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NMRR-19-3298-50711
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Caregiver Burden
Keywords: Informal caregiver of person with dementia; Educational intervention
MeSH Terms: conditions — Caregiver Burden | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receive normal care
- Intervention (Experimental): Educational intervention
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Educational module and video
  Arms: Intervention

SUMMARY:
The goal of this intervention study is to test whether the educational intervention work well or not on informal caregiver of person with dementia. The main question it aims to answer is does the educational intervention will help to reduce the caregiver burden experience by the informal caregiver.

Participants will be given an educational module and short videos that they can refer to gain more knowledge and skills in caring for the person with dementia.

DETAILED DESCRIPTION:
Caregivers for this study will be recruited at the geriatric, neurology and, psychiatry outpatient clinic. The caregiver will be approached by the primary researcher and explained about the details of the study. The caregivers will be given the participant information sheet and if they agree to participate in the study, written informed consent will be obtained.

The researcher will then check the eligibility of the caregiver to participate. If the caregiver was eligible to participate, they will be ask to provide contact details for researcher to assign tentative date for the virtual educational session. The caregiver will be then randomly assigned to control or intervention group before the baseline data were collected. This study will use equal allocation with a ratio of one to one for each two groups. The caregiver will be randomly allocated by using permuted block randomization technique. This study will be conducted as single blind study. Only the respondents would be blinded and concealed from the group allocation.

The intervention group will be given the educational intervention which are educational module and short videos related to dementia care. After the baseline data collection, the soft copy of the educational module will be shared to the participants via WhatsApp messenger so that they can review the module before the virtual educational session. One short educational video will be then shared to all the participants through individual WhatsApp in each Wednesday of the week for 12 weeks. Each of the short video will contain subtopics of the educational module and each video will be around two to three minutes. After the video shared to the participants, they are encouraged to ask any questions related to the content of the video.

ELIGIBILITY:
Inclusion Criteria:

1. Informal caregiver of person with dementia (children, children in law, grandchildren, grandchildren in law, spouses, siblings, parents).
2. Age 18 years old and above.
3. Able to understand, read and speak Bahasa Malaysia language

Exclusion Criteria:

1. Caregiver with previous history of mental illness.
2. Caregiver with physical disabilities that cause limitation in providing care for person with dementia.
3. Paid informal caregiver (maid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden | Baseline, 2 weeks after the end of educational intervention session, and 3 months after intervention
  The caregiver burden measured by using Zarit Burden Interview (ZBI). ZBI consisted of 22 items with all negative statements. The scoring will be zero for never, one for rarely, two for sometimes, three for quite frequently and four for nearly always. The scoring can be from zero to 88 with scoring of 0 to 21 little or no burden, 21 to 40 mild to moderate burden, 41 to 60 moderates to severe burden, and 61 to 88 severe burdens.

SECONDARY OUTCOMES:
Socio-demographic characteristic | Baseline
  To describe the characteristics (age, gender, ethnic, level of education, employment status, relationship with demented person, monthly household income) of the caregiver of person with dementia
Caregiving characteristics | Baseline
  To describe the caregiving characteristics (time spent with dementia person, severity of dementia person, functional abilities of dementia person, supports group availability) of the caregiver of person with dementia
Caregiver knowledge on dementia | Baseline, 2 weeks after the end of educational intervention session, and 3 months after intervention
  Caregiver knowledge on dementia will be based on the dementia knowledge assessment scale (DKAS) which use to explore what different individuals understand about dementia by using a multi-domain measure of dementia knowledge. The scale use five answer of measurement which is false, probably false, probably true, true and I do not know. Two points of score would be given for an answer of true to a true statement and false to a false statement. One point of score would be given for an answer of probably true to a true statement and probably false to a false statement. If the respondents give an answer of true on a false statement, false on a true statement and any answer of I do not know would be given zero point. The maximum score for the DKAS is 50 points and the respondent can be categorized on having a good knowledge if they score 40 and above, moderate level of knowledge if the score 25 to 39, and poor level of knowledge if they score below than 25 points.
Caregiver self-esteem | Baseline, 2 weeks after the end of educational intervention session, and 3 months after intervention
  The caregiver self-esteem will be measure by using the short sense of competence questionnaire. The scale is used to measure three domains which are the caregiver consequences of involvement in care for caregiver personal life, satisfaction with one's own performance as a caregiver and satisfaction with the demented person as a recipient care. The scoring for the scale would be one for strongly agree, two for agree, three for neutral, four for disagree and five for strongly disagree for the negative statement items. The scoring will be vice versa for the positive statement item. Higher scores indicate greater levels of competence.
Caregiver mastery | Baseline, 2 weeks after the end of educational intervention session, and 3 months after intervention
  The caregiver mastery is measured by using the Pearlin Mastery Scale by Pearlin and Schooler which used to explore protective buffer for caregiver' mental and physical health and well-being, when facing persistent life stresses, such as economic and occupational hardships.The scale used four-point Likert scale with one for strongly disagree, two for disagree, three for agree, and four for strongly agree. Items are summed, yielding a range from 7 to 28. Higher scores indicate greater levels of mastery.
Caregiver stress coping | Baseline, 2 weeks after the end of educational intervention session, and 3 months after intervention
  The caregiver stress coping will be measure by using The Coping Strategy Indicator (CSI) that is used to measures coping responses to a specific stressful event. Respondents who have high scored in the problem-solving scale were not likely to seek distraction or support. High score in the social support and avoidance scale indicates that, caregivers are not likely sought for information or distraction. High score in the avoidance subscale also most commonly predictive of negative mental health outcome such as depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nuraisyah Hani Zulkifley, Principal Investigator — Universiti Putra Malaysia